CLINICAL TRIAL: NCT00854399
Title: Screening and Identification of Novel Diagnostic and Prognostic Biomarkers on Ovarian Cancers
Brief Title: Screening and Identification of Ovarian Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Fang Cheng/Associate Professor, National Taiwan Unviersity Hospital
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200706002R
Record Dates: First submitted 2008-04-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Staging surgery or debulking surgery — Staging surgery or debulking surgery

SUMMARY:
Ovarian cancer is the first mortality rate of gynecologic malignancies. The incidence of ovarian cancer increased in recent 10 years and it has become the ninth cause of malignancies in the women in Taiwan. From the above-mentioned data, ovarian cancer indeed is a disease that should be respected, however, there were only few of research work focusing on it in Taiwan. Despite the widespread use of aggressive cytoreductive surgery and the introduction of chemotherapy regimens, the overall survival has changed little over the last two decades. The basic problem in treating epithelial ovarian cancer is that once it has spread beyond the ovary, it is exceedingly difficult to control and ultimately to cure. More than 70% of ovarian cancer patients were advanced stage when diagnosed. To study the mechanisms of carcinogenesis, progression, and metastasis of ovarian cancer will help us understand this disease and develop new treatment strategies for ovarian cancer in the future.

We have established an ascites-generating intraperitoneal tumor cell line-WF3 in the mouse model in our previous two-year project of NSC grant (grant number (NSC90-2314-B-002-457 and NSC91-2341-B-002-315). Our group found that, mesothelin, this molecule is highly related with the carcinogenesis, tumor progression and tumor metastasis in our animal model and human cancer tissues. To further evaluate the role of mesothelin in ovarian cancer and elucidate the potential of mesothelin as a target antigen for immunotherapy,

DETAILED DESCRIPTION:
Methods:

All of the patients received four to six courses of adjuvant platinum-containing chemotherapy. Histologic grading was according to International Union against Cancer criteria (28). The stage of disease was classified according to the International Federation of Gynecology and Obstetrics (FIGO, 1987). Pelvic and paraaortic lymph node samplings will be performed, if the disease will be confined to within the ovary or will be without a ruptured capsule. The histopathologic data, including histologic type and histologic grade, will be evaluated by a certified pathologist. The maximal diameter of the residual tumor after surgery will be also recorded. All patients will be followed up at 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian carcinoma who undergo hysterectomy, bilateral oophorectomy and tubal resection, omentectomy, and appendectomy will be enrolled and the clinical data will be obtained from our hospital.

Exclusion Criteria:

* None

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-01; Primary Completion 2006-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | from disease diagnosis to death

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YL, Lin HW, Chien CL, Lai YL, Sun WZ, Chen CA, Cheng WF. BTLA blockade enhances Cancer therapy by inhibiting IL-6/IL-10-induced CD19high B lymphocytes. J Immunother Cancer. 2019 Nov 21;7(1):313. doi: 10.1186/s40425-019-0744-4. PMID 31753019